CLINICAL TRIAL: NCT06866977
Title: A Single-arm, Open-label Clinical Study to Evaluate the Efficacy and Safety of VRT106 in Combination With Chemotherapy for Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-C04
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: Advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRT106 combination with chemotherapy (Experimental): VRT106 combination with chemotherapy
  Interventions: Drug: Oncolytic virus VRT106; Drug: Chemotherapy

INTERVENTIONS:
Drug: Oncolytic virus VRT106 — VRT106, IV
  Other Names: VRT106
Drug: Chemotherapy — 21 days/cycle

SUMMARY:
This is a single-center, single-arm, open label investigator-initiated clinical study to evaluate the efficacy and safety of VRT106 in combination with chemotherapy in the treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open label investigator-initiated clinical study to evaluate the efficacy and safety of VRT106 in combination with chemotherapy in the treatment of advanced pancreatic cancer.

The study is planned to enroll 10 subjects. The entire study consists of a screening period of up to 28 days, treatment period, and a follow-up period (safety follow-up 28 days after the final study dose and survival follow-up once every 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an Institutional Review Board -approved informed consent prior to performing any of the Screening Visit procedures.
* Males and females≥18 years of age, inclusive, at the Screening Visit.
* Have unresectable pancreatic cancer as determined by imaging or surgical exploration and locally advanced or metastatic pancreatic ductal adenocarcinoma (including adenosquamous carcinoma) as confirmed by histology or cytology.
* No prior systemic therapy for unresectable locally advanced and metastatic pancreatic cancer.
* Have at least one measurable lesion according to RECIST v1.1 criteria.
* An Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
* Expected survival time of≥3 months.
* No serious hematologic and cardiac abnormalities of the liver, kidneys, or coagulation functions.

Exclusion Criteria:

* Have suffered from other malignant tumors in the past 5 years, except for cured basal cell skin cancer, non-melanoma skin cancer, and cervical cancer in situ.
* Previous treatment with other oncolytic viruses.
* Immunocompromised patients.
* Known alcohol or drug dependency.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-12 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | About 3 years
  Incidence rate of TRAE

SECONDARY OUTCOMES:
Overall survival rate | About 3 years
  Overall survival rates at 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China